CLINICAL TRIAL: NCT00370773
Title: Treatment of Chronic Low Back Pain With Spinal Cord Stimulation: Comparison of Subthreshold Intraspinal Nerve Root Stimulation With Subthreshold and Suprathreshold Dorsal Column Stimulation and a Secondary Study of the Effect of Pulse Width
Brief Title: Comparison of Intraspinal Nerve Root Stimulation With Dorsal Column Stimulation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Enrolling
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Lyn Pimentel, Clinical Project Manager, Boston Scientific Corporation
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: SCS0705
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-08

CONDITIONS: Back Pain
Keywords: Failed Back Surgery Syndrome; Back Pain; Chronic Pain; Spinal Cord Stimulation
MeSH Terms: conditions — Back Pain; Failed Back Surgery Syndrome; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Precision Spinal Cord Stimulation System

SUMMARY:
This study will systematically evaluate the programming parameters of the Precision Spinal Cord Stimulation Device to optimally relieve pain while minimizing any uncomfortable side effects.

DETAILED DESCRIPTION:
This study will investigate the efficacy of subthreshold intraspinal nerve root stimulation (INRS) in treating back pain. The efficacy of this strategy will be tested against dorsal column stimulation (DCS), the commonly-accepted technique for spinal cord stimulation. DCS will be tested at subthreshold and suprathreshold (perceptible) amplitudes. A substudy will involve patients who prefer suprathreshold DCS over INRS and subthreshold DCS. Its purpose is to systematically assess the pain relief afforded by a number of programs with different pulse widths. The overall purpose of this study is to investigate methods of making pain relief via electrical stimulation more comfortable by either using subthreshold amplitudes or by adjusting the pulse width of perceptible stimulation to a more pleasing range.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic low back pain following spine surgery (Failed Back Surgery Syndrome.
* Be an appropriate candidate for Spinal Cord Stimulation (SCS) and for the surgical procedures required for SCS.
* Have experienced significant though short-lived pain relief with local anesthetic injection.
* Be 18 years of age or older.
* Be willing and able to comply with all study related procedures and visits.
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have any significant medical condition that is likely to interfere with study procedures.
* Have any evidence of neurologic instability.
* Have any other chronic pain condition.
* Have a condition currently requiring or likely to require the use of MRI or diathermy.
* Have an active implantable device.
* Are pregnant or planning to become pregnant in the next year.
* Are a current substance abuser (including alcohol and illicit drugs).
* Have a significant psychiatric disorder.
* Have participated in any drug or device trial in the last 4 weeks or plan to participate in any other trial during the duration of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare subthreshold intraspinal nerve root stimulation (INRS) with subthreshold and suprathreshold dorsal column stimulation (DCS). | 1 year
The primary safety endpoint is incidence of adverse events. | Throughout Study

SECONDARY OUTCOMES:
The secondary objectives of this study are to assess the effect of different stimulation types on average pain and pain-related disability, and to assess the subjective comfort of paresthesia with different pulse widths. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yearwood, MD, Principal Investigator — Comprehensive Pain and Rehabilitation
Locations (1):
- Comprehensive Pain & Rehabilitation, Daphne, Alabama, United States